CLINICAL TRIAL: NCT05781347
Title: Endoscopic Treatment of Gastro-esophageal Reflux Disease with Application of Radiofrequency Energy to the Lower Esophageal Sphincter (Stretta) Versus Conservative Treatment, Prospective Randomized Study
Brief Title: Stretta Versus Conservative Treatment
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Military University Hospital, Prague (Other)
Responsible Party: Principal Investigator, Katerina Kostalova, MD, Principal Investigator, Military University Hospital, Prague
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 108/17-12/2022
Record Dates: First submitted 2023-02-16; First posted 2023-03-23 (Actual); Last update posted 2025-01-07 (Actual); Status verified 2025-01

CONDITIONS: GERD
MeSH Terms: conditions — Gastroesophageal Reflux

STUDY DESIGN:
Intervention Model Description: Patients will be randomized (ratio 1:1) into two groups: one receiving the Stretta therapy and the other undergoing conservative treatment with proton pump inhibitors (PPIs). The initial plan to stratify patients into obese and non-obese groups was revised due to recruitment challenges. The study now includes all eligible patients with gastroesophageal reflux disease (GERD), regardless of body weight, provided they meet the inclusion criteria.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Patients receiving Stretta (Active Comparator)
  Interventions: Procedure: Radiofrequency Energy to the LES (Stretta Procedure); Device: Stretta
- Patients receiving Conservative therapy/PPI (No Intervention)

INTERVENTIONS:
Procedure: Radiofrequency Energy to the LES (Stretta Procedure) — The Stretta procedure is an endoscopic treatment performed under general anesthesia. It utilizes radiofrequency (RF) energy delivered to the lower esophageal sphincter (LES) and the gastric cardia to enhance the antireflux barrier.
  Arms: Patients receiving Stretta
Device: Stretta — Stretta is a FDA approved device for the management of GERD.
  Arms: Patients receiving Stretta

SUMMARY:
Gastroesophageal reflux disease (GERD) is one of the most common diseases of the gastrointestinal tract. Obesity is a significant risk factor for GERD; however, treatment outcomes in obese patients remain challenging. In the Czech Republic, therapeutic options are currently limited to conservative treatment, including pharmacotherapy and lifestyle modifications, or surgical interventions, both of which have known limitations. Stretta is a minimally invasive endoscopic therapy using radiofrequency energy delivered to the esophagogastric junction (EGJ) and cardia, aimed at enhancing the antireflux barrier.

This study evaluates the effectiveness and safety of the Stretta procedure compared to conservative treatment in managing GERD. Initially designed to compare outcomes between obese and non-obese populations, the study was expanded to include all GERD patients due to recruitment challenges and the need to meet strict eligibility criteria. These criteria ensure reliable results by focusing on patients with confirmed pathological GERD while excluding those with hiatal hernias ≥ 2 cm, severe esophagitis, or functional esophageal disorders such as hypersensitivity. The study aims to provide comprehensive data on the use of Stretta in the Czech Republic and its role in GERD management.

DETAILED DESCRIPTION:
Gastroesophageal reflux disease (GERD) is a significant clinical issue that substantially impairs patients' quality of life. Chronic symptoms such as heartburn, regurgitation, and chest pain, along with extraesophageal manifestations (e.g., laryngopharyngeal reflux), often drive patients-especially younger individuals-to seek effective treatment options. Many of these patients are motivated by the desire to reduce or eliminate long-term proton pump inhibitor (PPI) use, given concerns about potential side effects and dependence on medication.

The Stretta procedure, a minimally invasive endoscopic therapy using radiofrequency energy delivered to the esophagogastric junction (EGJ) and cardia, has shown promise in addressing these concerns by enhancing the antireflux barrier. This study aims to evaluate the effectiveness and safety of Stretta compared to conservative treatment in improving GERD management in the Czech Republic.

Initially, the study was designed to compare outcomes between obese and non-obese populations. However, due to recruitment challenges and the need for strict inclusion criteria, it was expanded to include all patients with confirmed pathological GERD. Participants are carefully selected based on stringent eligibility criteria, including pathological GERD confirmed by 24-hour pH-metry with impedance and exclusion of those with hiatal hernias ≥ 2 cm, severe esophagitis, or functional esophageal disorders such as esophageal hypersensitivity.

The primary goal of this study is to improve patients' quality of life and reduce the reliance on chronic PPI therapy. Secondary objectives include assessing the safety profile of the Stretta procedure and its effectiveness compared to conservative management in a broader GERD population. By focusing on these outcomes, the study seeks to provide valuable insights into the role of Stretta as a therapeutic option in GERD management and its potential to fill a critical gap in current treatment modalities.

ELIGIBILITY:
Inclusion Criteria:

Verified symptomatic GERD despite PPI use, with persistent symptoms, desire to discontinue PPIs, or intolerance to them.

Pathological gastroesophageal reflux confirmed by positive 24-hour pH-metry with impedance.

Normal findings on high-resolution esophageal manometry (HRM) according to CCv4.0.

Age ≥ 18 years. Signed informed consent for participation in the trial and invasive procedures.

Exclusion Criteria:

Active severe reflux esophagitis (Los Angeles classification grade C or D). Barrett's esophagus. Esophageal peptic stricture or eosinophilic esophagitis. Hiatal hernia ≥ 2 cm. Malignancies. Abnormal findings on high-resolution esophageal manometry. Esophageal or subcardial varices. Pregnancy. Severe comorbidities or increased perioperative risk. Age > 70 years due to increased perioperative risk and common comorbidities. Symptoms primarily attributable to functional dyspepsia, significant anxiety, or depression, with overlap to other disorders of gut-brain interaction (DGBI).

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2022-09-01 (Actual); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Proton pump inhibitors (PPI) use | 6 months
  Cessation or reducing the dose of PPI by at least 50% from baseline
Proton pump inhibitors (PPI) use | 12 months
  Cessation or reducing the dose of PPI by at least 50% from baseline
GERD Health Related Quality of Life questionaire | 6 months
  Change in symptom severity assessed by validated reflux questionnaire
GERD Health Related Quality of Life questionaire | 12 months
  Change in symptom severity assessed by validated reflux questionnaire (GERD - HRQL)
Reflux Severity Index score | 6 months
  Change in symptom severity assessed by validated reflux questionnaire
Reflux Severity Index score | 12 months
  Change in symptom severity assessed by validated reflux questionnaire

SECONDARY OUTCOMES:
24h pH-metry with impedance | 6 months
  Change in pH-metric parameters (Acid Exposure Time - AET)
24h pH-metry with impedance | 12 months
  Change in pH-metric parameters (Acid Exposure Time - AET)

CONTACTS AND LOCATIONS:
Locations (1):
- Military University Hospital Prague, Prague, Czechia

IPD SHARING:
Plan to Share IPD: No